CLINICAL TRIAL: NCT03636893
Title: Dragon III- Phase 2: The Preliminary Efficacy Study of FLOT Versus SOX Regimen as Neoadjuvant Chemotherapy for Patients With Locally Advanced Gastric Cancer: Open-label, Randomized Controlled Trial
Brief Title: Dragon III: Neoadjuvant Chemotherapy (FLOT Versus SOX) for Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, BIRENDRA KUMAR SAH, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dragon III
Record Dates: First submitted 2018-08-01; First posted 2018-08-17 (Actual); Results first posted 2020-06-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; Chemotherapy Effect
Keywords: Neoadjuvant chemotherapy; perioperative chemotherapy; Systemic chemotherapy; FLOT; SOX; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomly assigned(1:1) either to FLOT or SOX group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLOT Chemotherapy regimen (Experimental): A total of four preoperative and four postoperative cycles of FLOT chemotherapy administered
  A cycle consists of Day 1 5-fluorouracil(5-FU) 2600mg/M2 administered via an intravenous peripherally inserted central venous catheter(PICC) for 24 hour Leucovorin 200mg/M2 intravenous Oxaliplatin 85mg/ M2 intravenous Docetaxel 50mg/M2 intravenous
  Repeated every 15th day
  Interventions: Drug: FLOT Chemotherapy
- SOX Chemotherapy regimen (Active Comparator): Three preoperative cycles and three postoperative cycles of SOX chemotherapy administered
  A cycle consist of Day 1: Oxaliplatin 130mg/M2 intravenous Day 1-14 Tegafur gimeracil oteracil potassium capsule 80mg/M2 oral (twice daily)
  Repeated every 21st day
  Interventions: Drug: SOX Chemotherapy

INTERVENTIONS:
Drug: FLOT Chemotherapy — 5-FU+Leucovorin+Docetaxel+Oxaliplatin
  Other Names: FLOT
  Arms: FLOT Chemotherapy regimen
Drug: SOX Chemotherapy — Oxaliplatin+Tegafur gimeracil oteracil potassium capsule (TGO)
  Other Names: SOX
  Arms: SOX Chemotherapy regimen

SUMMARY:
Safety and efficacy study of neoadjuvant chemotherapy (FLOT versus SOX) for gastric cancer patients in high volume center of China

DETAILED DESCRIPTION:
DRAGON III research, Neoadjuvant Chemotherapy (FLOT versus SOX) for Gastric Cancer, is an investigator initiated; phase II, open label, randomised controlled study. This study will be conducted and analyzed by the Gastrointestinal department（Unit III）of the Ruijin Hospital and the project is supported by the Institute of Digestive Surgery, Shanghai, which is a state key research center. This study will be monitored by the Clinical Research Center of the Ruijin hospital (Official body which is responsible to guide and monitor all types of research at Ruijin hospital). Primary endpoint and secondary endpoint is described above. The aim of this study to obtain preliminary result and further conduct a large scale multi-center randomised controlled trial(RCT) study.

ELIGIBILITY:
Inclusion criteria:

* Histology confirmed non-obstructive adenocarcinoma of the stomach or esophagogastric junction.
* Clinical stage: cTNM: stage III or above
* Performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2 (normal to symptomatic but in bed less than half the day)
* Clinically fit for systemic chemotherapy and gastric cancer surgery, i.e. adequate renal, hepatic, hematologic, and pulmonary function.
* Written informed consent

Exclusion criteria:

* Clinically unfit for systemic chemotherapy and gastric cancer surgery, i.e. uncontrolled cardiac disease, or other clinically significant uncontrolled comorbidities, unable to undergo general anesthesia
* Confirmed distant metastases
* Locally advanced inoperable disease (Clinical assessment)
* Relapse of gastric cancer
* Malignant secondary disease
* Prior chemo or radiotherapy
* Inclusion in another clinical trial
* Known contraindications or hypersensitivity for planned chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2025-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birendra Kumar Sah, PH D, Principal Investigator — Ruijin Hospital; Chen Li, PH D, Study Director — Ruijin Hospital; Zhenggang Zhu, PH D, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sah BK, Yu Z, Zhang B, Yuan F, Zhang H, Li J, Ma T, Shi M, Zhu Z, Zheng Y, Liu W, Yan C, Li C, Zhu Z. Neoadjuvant FLOT versus SOX chemotherapy in locally advanced gastric cancer: secondary outcomes of a single-centre, open-label, randomised, exploratory phase 2 trial. EClinicalMedicine. 2025 Oct 5;88:103494. doi: 10.1016/j.eclinm.2025.103494. eCollection 2025 Oct. PMID 41181842
- [Derived] Sah BK, Zhang B, Zhang H, Li J, Yuan F, Ma T, Shi M, Xu W, Zhu Z, Liu W, Yan C, Li C, Liu B, Yan M, Zhu Z. Neoadjuvant FLOT versus SOX phase II randomized clinical trial for patients with locally advanced gastric cancer. Nat Commun. 2020 Nov 30;11(1):6093. doi: 10.1038/s41467-020-19965-6. PMID 33257672

RESULTS

PARTICIPANT FLOW:
Groups:
- FLOT Chemotherpy Regimen: A total of four preoperative and four postoperative cycles of FLOT chemotherapy administered
  A cycle consists of Day 1 5-fluorouracil (5-FU) 2600mg/M2 administered via an intravenous peripherally inserted central venous catheter (PICC) for 24 hour Leucovorin 200mg/M2 intravenous Oxaliplatin 85mg/ M2 intravenous Docetaxel 50mg/M2 intravenous
  Repeated every 15th day
  Three drug Chemotherapy: 5-FU+Leucovorin+Docetaxel+Oxaliplatin
- SOX Chemotherapy Regimen: Three preoperative cycles and three postoperative cycles of SOX chemotherapy administered
  A cycle consists of Day 1: Oxaliplatin 130mg/M2 intravenous Day 1-14 Tegafur gimeracil oteracil (TGO) potassium capsule 80mg/M2 oral (twice daily)
  Repeated every 21st day
  Two drug Chemotherapy: Oxaliplatin+TGO
Period: Overall Study
Arm/Group | FLOT Chemotherpy Regimen | SOX Chemotherapy Regimen
Started | 40 | 34
Completed | 31 | 24
Not Completed | 9 | 10
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Refusal to surgery | 4 | 3
Not completed — Early surgery (for acute bleeding) | 3 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol(PP) population
Groups:
- FLOT Chemotherpy Regimen: A total of four preoperative and four postoperative cycles of FLOT chemotherapy administered
  A cycle consists of Day 1 5-FU 2600mg/M2 administered via intravenous PICC for 24 hour Leucovorin 200mg/M2 intravenous Oxaliplatin 85mg/ M2 intravenous Docetaxel 50mg/M2 intravenous
  Repeated every 15th day
  Three drug Chemotherapy: 5-FU+Leucovorin+Docetaxel+Oxaliplatin
- Total: Total of all reporting groups
Arm/Group | FLOT Chemotherpy Regimen | SOX Chemotherapy Regimen | Total
Number analyzed (Participants) | 31 | 24 | 55
Age, Customized [Count of Participants; unit: Participants]
  <=60 | 7 | 14 | 21
  61-70 | 16 | 7 | 23
  71-80 | 8 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 22 | 14 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 24 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 31 | 24 | 55
BMI [Median (Full Range); unit: kg/m^2] | 23.56 [15.69 to 29.48] | 23.49 [17.31 to 27.82] | 23.56 [15.69 to 29.48]

OUTCOME MEASURES:

1. Primary Outcome: Total Percentage of Patients With Pathological Complete Tumor Regression (TRG1a) and Sub-total Tumor Regression (TRG1b) in the Primary Tumour
Description: Tumor regression grade (TRG), Becker criteria Grade 1a :Complete tumor regression: 0% residual tumor per tumor bed Grade 1b: Subtotal tumor regression: <10% residual tumor per tumor bed Grade 2: Partial tumor regression: 10-50% residual tumor per tumor bed Grade 3: Minimal or no tumor regression: >50% residual tumor per tumor bed
Time Frame: Three months
Population: Intention-to-treat (ITT) population
Measure: Count of Participants; unit: Participants
Groups:
- FLOT Chemotherpy Regimen: A total of four preoperative and four postoperative cycles of FLOT chemotherapy administered
  A cycle consist of Day 1 5-FU 2600mg/M2 administered via intravenous PICC for 24 hour Leucovorin 200mg/M2 intravenous Oxaliplatin 85mg/ M2 intravenous Docetaxel 50mg/M2 intravenous
  Repeated every 15th day
  Three drug Chemotherapy: 5-FU+CF+Docetaxel+Oxaliplatin
- SOX Chemotherapy Regimen: Three preoperative cycles and three postoperative cycles of SOX chemotherapy administered
  A cycle consist of Day 1: Oxaliplatin 130mg/M2 intravenous Day 1-14Tegafur gimeracil oteracil potassium capsule 80mg/M2 oral (twice daily)
  Repeated every 21st day
  Two drug Chemotherapy: Oxaliplatin+TGO
Arm/Group | FLOT Chemotherpy Regimen | SOX Chemotherapy Regimen
Number analyzed (Participants) | 40 | 34
Participants
  Grade 1a: Complete tumor regression | 1 | 0
  Grade 1b: Subtotal tumor regression | 7 | 11
  Grade 2: Partial tumor regression | 13 | 7
  Grade 3: Minimal or no tumor regression | 10 | 6
  Pathology not available | 9 | 10

2. Secondary Outcome: Disease-free Survival (DFS)
Description: Time from randomization to the first occurrence of local recurrence, regional recurrence, distant metastases, or death from any cause.
  Disease recurrence was assessed using CT imaging with contrast, upper endoscopy for local recurrence, histological confirmation when feasible, and multidisciplinary team review of imaging findings.
Time Frame: From randomization through 5 years follow-up (median follow-up 65.7 months)
Population: Intention-to-treat population including all 74 randomized patients regardless of treatment completion or protocol adherence. Complete vital status obtained for all patients with median follow-up of 65.7 months.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- FLOT Chemotherapy Regimen: A total of four preoperative and four postoperative cycles of FLOT chemotherapy administered
  A cycle consists of Day 1 5-fluorouracil(5-FU) 2600mg/M2 administered via an intravenous peripherally inserted central venous catheter(PICC) for 24 hour Leucovorin 200mg/M2 intravenous Oxaliplatin 85mg/ M2 intravenous Docetaxel 50mg/M2 intravenous
  Repeated every 15th day
  FLOT Chemotherapy: 5-FU+Leucovorin+Docetaxel+Oxaliplatin
- SOX Chemotherapy Regimen: Three preoperative cycles and three postoperative cycles of SOX chemotherapy administered
  A cycle consist of Day 1: Oxaliplatin 130mg/M2 intravenous Day 1-14 Tegafur gimeracil oteracil potassium capsule 80mg/M2 oral (twice daily)
  Repeated every 21st day
  SOX Chemotherapy: Oxaliplatin+Tegafur gimeracil oteracil potassium capsule (TGO)
Arm/Group | FLOT Chemotherapy Regimen | SOX Chemotherapy Regimen
Number analyzed (Participants) | 40 | 34
months | 23.0 [8.0 to 38.0] | 25.5 [12.0 to 38.9]
Statistical Analysis 1: Comparison: FLOT Chemotherapy Regimen vs SOX Chemotherapy Regimen; Disease-free survival analysis in intention-to-treat population. DFS defined as time from randomization to first occurrence of local recurrence, regional recurrence, distant metastases, or death from any cause; Test type: Other — Two-sided log-rank test comparing disease-free survival between treatment groups. No adjustment for multiple comparisons as this was a pre-specified secondary endpoint. Statistical significance set at P <0.05; p = 0.842, Log Rank — P-value from two-sided log-rank test. Alpha level set at 0.05; Kaplan-Meier survival analysis with log-rank test for between-group comparison. Analysis performed using SPSS version 30.0; Hazard Ratio (HR) = 1.060, 95% CI 2-sided [0.597 to 1.884] — Hazard ratio from Cox proportional hazards regression with FLOT as reference group; Kaplan-Meier method used to estimate DFS curves. Cox regression performed to calculate hazard ratios

3. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to death from any cause. Patients alive at the time of analysis were censored on the date of the last follow-up visit. Vital status was verified through multiple sources: direct clinical follow-up, telephone contact, cross-referencing with local death registry records, and review of medical records from other healthcare facilities.
Time Frame: From randomization through 5 years follow-up (median follow-up 65.7 months)
Population: Intention-to-treat population including all 74 randomized patients regardless of treatment completion or protocol adherence. Complete vital status obtained for all patients. At data cut-off, 41 deaths occurred: 21 (52.5%) in FLOT group and 20 (58.8%) in SOX group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FLOT Chemotherapy Regimen | SOX Chemotherapy Regimen
Number analyzed (Participants) | 40 | 34
months | 61.5 [61.5 to NA] — Upper CI limit not estimable - median survival not reached due to >50% of FLOT patients remaining alive at data cutoff. | 67.8 [25.7 to 109.9]
Statistical Analysis 1: Comparison: FLOT Chemotherapy Regimen vs SOX Chemotherapy Regimen; Primary survival analysis comparing overall survival between neoadjuvant FLOT and SOX regimens in intention-to-treat population; Test type: Other — Two-sided log-rank test comparing overall survival between treatment groups. No adjustment for multiple comparisons as this was a pre-specified secondary endpoint. Statistical significance set at P <0.05; p = 0.759, Log Rank — P-value from two-sided log-rank test. No adjustment for multiple comparisons as overall survival was a pre-specified secondary endpoint. Alpha level set at 0.05; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.101, 95% CI 2-sided [0.595 to 2.036] — Hazard ratio from Cox proportional hazards regression with FLOT as reference group; Kaplan-Meier method used to estimate survival curves. Cox regression performed to calculate hazard ratios. Multivariable analysis performed to identify independent predictors

ADVERSE EVENTS:
Time Frame: From randomization through 5 years follow-up (median follow-up 65.7 months)
Description: All 74 randomized participants were assessed for all-cause mortality per intention-to-treat analysis. According to the study protocol, serious adverse events and other adverse events were systematically collected for all 74 participants during the study period, including events leading to treatment discontinuation. Adverse events leading to dropout were captured as protocol violations or serious adverse events as appropriate.
Arm/Group | FLOT Chemotherpy Regimen | SOX Chemotherapy Regimen
All-Cause Mortality (participants affected / at risk) | 21/40 | 20/34
Serious Adverse Events (participants affected / at risk) | 9/40 | 8/34
Other Adverse Events (participants affected / at risk) | 9/40 | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLOT Chemotherpy Regimen (N=40) | SOX Chemotherapy Regimen (N=34)
Overall postoperative complication (Surgical and medical procedures) | 9 | 8
Postoperative complications: Death (Surgical and medical procedures) | 0 | 0
Grade IV hematological toxicity with multiple organ failure (Blood and lymphatic system disorders) | 0 | 1 — Grade IV hematological toxicity with multiple organ failure
Acute cerebral infarction (Nervous system disorders) | 1 | 0 — Acute cerebral infarction
Deep venous thrombosis (Vascular disorders) | 0 | 1 — Deep venous thrombosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLOT Chemotherpy Regimen (N=40) | SOX Chemotherapy Regimen (N=34)
Grade 3+Grade 4 Decrease in white blood cells (Blood and lymphatic system disorders) | 1 | 0 — Common Terminology Criteria for Adverse Events (CTCAE)Version 4.0: Decrease in white blood cells
Grade 3+Grade 4 Neutrophil count decreased (Blood and lymphatic system disorders) | 2 | 2
Grade 3+Grade 4 Platelet count decreased (Blood and lymphatic system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
ALT (Hepatobiliary disorders) | 0 | 0
AST (Hepatobiliary disorders) | 1 | 0
Acute bleeding requiring emergency surgery (Gastrointestinal disorders) | 3 | 0 — Acute bleeding requiring emergency surgery

LIMITATIONS AND CAVEATS:
This is a preliminary result of phase II study with inadequate sample numbers. A phase III multi center randomised controlled trial is necessary to justify these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT03636893/Prot_SAP_000.pdf